CLINICAL TRIAL: NCT01287169
Title: BPA Biomonitoring Study in Cashiers
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911074; 11-E-N074
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2012-12-04

CONDITIONS: Bisphenol A
Keywords: Bisphenol A

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
We intend to conduct a pilot study designed to measure BPA levels before and after occupational exposure to thermal paper used in cash registers. We will recruit cashiers from a local commercial store that is currently still using BPA-laden thermal paper and plans to switch to BPA-free paper in the near future. The study uses a within-subject comparison design, using serum and urine samples to determine whether BPA is detectable in the study population at sufficient levels to measure differences in paired samples. Two phases of sample collection are proposed: Phase I - collecting paired samples on two separate occasions before the implementation of BPA-free thermal paper use in cash registers; and Phase II - collecting paired samples on two separate occasions after the implementation of this change in thermal paper.

...

DETAILED DESCRIPTION:
We intend to conduct a pilot study designed to measure BPA levels before and after occupational exposure to thermal paper used in cash registers. We will recruit cashiers from a local commercial store that is currently still using BPA-laden thermal paper and plans to switch to BPA-free paper in the near future. The study uses a within-subject comparison design, using serum and urine samples to determine whether BPA is detectable in the study population at sufficient levels to measure differences in paired samples. Two phases of sample collection are proposed: Phase I - collecting paired samples on two separate occasions before the implementation of BPA-free thermal paper use in cash registers; and Phase II - collecting paired samples on two separate occasions after the implementation of this change in thermal paper.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female 18 years of age or older at the time of enrollment
* Employed as a cashier at the site location
* Anticipate continued employment at this business for the duration of both phases of the study
* Able to understand and provide written informed consent to participate in the study
* Have a minimum of 24 hours off from work before providing pre-shift samples
* Participants may be healthy or have preexisting conditions.

Field Site Inclusion Criteria:

* Have a minimum of 20 employed cashiers
* Use BPA-laden thermal paper and is planning to switch to BPA-free thermal paper
* Have a private area that the study nurse can use for enrollment and collection of biological samples
* Willing to collaborate with study team to conduct study on-site

EXCLUSION CRITERIA:

-There are no additional exclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01-10; Study Completion 2012-12-04

CONTACTS AND LOCATIONS:
Overall Officials: John Bucher, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)

REFERENCES:
- [Background] Biedermann S, Tschudin P, Grob K. Transfer of bisphenol A from thermal printer paper to the skin. Anal Bioanal Chem. 2010 Sep;398(1):571-6. doi: 10.1007/s00216-010-3936-9. Epub 2010 Jul 11. PMID 20623271
- [Background] Calafat AM, Ye X, Wong LY, Reidy JA, Needham LL. Exposure of the U.S. population to bisphenol A and 4-tertiary-octylphenol: 2003-2004. Environ Health Perspect. 2008 Jan;116(1):39-44. doi: 10.1289/ehp.10753. PMID 18197297
- [Background] Kang JH, Kondo F, Katayama Y. Human exposure to bisphenol A. Toxicology. 2006 Sep 21;226(2-3):79-89. doi: 10.1016/j.tox.2006.06.009. Epub 2006 Jun 16. PMID 16860916